CLINICAL TRIAL: NCT05790226
Title: A Prospective Pre-Market Proof-of-Concept Study for Ex Vivo Raman Spectroscopy Measurements on Excised Lung Tissue With the Sentry System
Brief Title: Sentry Study: Raman Spectroscopy on Ex Vivo Lungs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor stopped study
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Sentry-2000-CIP-003
Record Dates: First submitted 2023-01-25; First posted 2023-03-30 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Raman Spectroscopy (Experimental): Acquiring Raman spectroscopy data points ex vivo on recently excised lung tissue
  Interventions: Device: Sentry System

INTERVENTIONS:
Device: Sentry System — any labelling or contrast agents. The Sentry System uses the Sentry Probe, a flexible cable that terminates in a stylus that delivers a small beam of light to the surface of the excised tissue specimen and collects the Raman spectrum of the light coming back from the same area of the specimen.

SUMMARY:
In this proof-of-concept, ex vivo study, the study team will investigate whether Raman spectroscopy technology is a good candidate for the identification of cancerous lung tissue.

DETAILED DESCRIPTION:
Lung cancer is the most prevalent form of cancer worldwide and the leading cause of cancer-related deaths. Despite recent advances in treatment, the five-year survival rate remains below 25% [State of Lung Cancer Report 2021,American Lung Association. This is largely due to the fact that most patients are diagnosed only at advanced stages of the disease when treatments are ineffective and the prognosis is poor. The National Lung Screening Trial demonstrated the utility of lung cancer screening by low-dose computed tomography (CT) to improve early detection\ and reduce lung cancer-related mortality by 20%. Earlier detection of lung lesions in turn created an increased need for better early diagnosis modalities.

Reveal Surgical is developing medical devices for tissue characterization based on Raman spectroscopy technology.

In this proof-of-concept, ex vivo study, the study team will investigate whether Raman spectroscopy technology is a good candidate for the identification of cancerous lung tissue.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above,
* With suspected or confirmed diagnosis of lung cancer,
* Scheduled for lobectomy surgery,
* Able to give informed consent.

Exclusion Criteria:

* Suspected or confirmed diagnosis of mucinous adenocarcinoma of the lung
* Undergoing neoadjuvant therapy. (This exclusion criterion is intended to minimize confounding optical signals such as fluorescence or near-infrared Raman signals that could arise from the presence of chromophores derived from neoadjuvant medication.)
* Previously diagnosed with cystic fibrosis or other lung disease, with the exception of Chronic Obstructive Pulmonary Disease (COPD) and ILD (Interstitial Lung Disease), i.e., patients with COPD or ILD will not be excluded from the study.
* Tumor size below 1cm3
* Resected lobe does not allow Surgical Pathology team to section two study specimens of minimal size 1.5cm × 1.5cm. In this case the patient will be found ineligible after consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
investigate the variability of the Raman spectra using data points ex vivo on recently excised lung tissue, with at least one third of spectra labeled as normal and cancerous based on subsequent histopathology assessment. | 1 year
  whether ex vivo cancerous and normal human lung tissue yield distinct Raman signatures.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No